CLINICAL TRIAL: NCT06600828
Title: Study's Care of Acute Pancreatitis at Saint-Etienne University Hospital.
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN902024/CHUSTE
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Acute Pancreatitis
Keywords: Internal Medicine Unit efficiency; Retrospective observational study; Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Internal Medicine Unit arm: It includes all patients hospitalized in the Internal Medicine Unit. Patients may have been previously hospitalized in the emergency department or in another department such as intensive care.
  Interventions: Other: Data collection
- The hepato-gastro-enterology Unit arm: It includes all patients hospitalized in the Gastroenterology unit. Patients may have been previously hospitalized in the emergency department or in another department such as intensive care.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collected: Socio-demographic, hospital, clinical, biological, and imaging data

SUMMARY:
Internal medicine units treat patients with undifferentiated or multisystem diseases, with a non-specific organ approach.

In some cases, patients with single-organ disease may be admitted to internal medicine wards. Acute pancreatitis is the most common gastrointestinal illness requiring acute admission to hospital. It is characterised by local and systemic inflammation of the pancreas corresponding to single-organ disease.

For patients with single-organ disease such as acute pancreatitis, it is not known whether admission to internal medicine is as effective as admission to a unit specialising in a specific organ, such as hepato-gastro-enterology.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* primary diagnosis of acute pancreatitis in Internal Medicine and gastroenterology.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients hospitalized from January 1, 2022, to December 31, 2023 in the University Hospital of Saint Etienne with a primary diagnosis of acute pancreatitis in Internal Medicine and gastroenterology will be included.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Performance Stay Length Index | From the date of inclusion to the date of discharge from hospital, assessed for up to 100 months
  "Performance Stay Length Index", is a measure used to evaluate the efficiency of hospital care in terms of patients' length of stay. This index is calculated by comparing the average length of stay of patients in a given service to a predefined reference, often based on established standards or goals.

SECONDARY OUTCOMES:
Rate of complications at 1 year | During one year from diagnosis
  Number of complications documented in the computerized medical record, one year from diagnosis.
Rate of rehospitalization at 1 year | During one year from diagnosis
  Number of hospitalizations documented in the computerized medical record, one year from diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kyria REGALADE, resident, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No